CLINICAL TRIAL: NCT07124806
Title: Comparison of Effectiveness of Two Techniques to Guide the Injection of Botulinum Toxin to Improve Gait in Post-stroke Patients: Randomized Clinical Trial
Brief Title: Comparison of Two Botox Injection Techniques to Improve Gait
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de los Andes, Chile (Other)
Collaborators: Fondo Nacional de Desarrollo Científico y Tecnológico, Chile (Other Government); Instituto Nacional de Rehabilitación Pedro Aguirre Cerda (Unknown)
Responsible Party: Principal Investigator, RODRIGO AANTONIO GUZMAN, PT, PhD, Universidad de los Andes, Chile
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: UAndes
Record Dates: First submitted 2025-08-08; First posted 2025-08-15 (Actual); Last update posted 2025-08-15 (Actual); Status verified 2025-08

CONDITIONS: Muscle Spasticity; Stroke Sequelae; Spasticity as Sequela of Stroke; Gait Disorders, Neurologic
Keywords: Post-Stroke; Gait analysis; Botulinum toxin; High-density electromyography
MeSH Terms: conditions — Muscle Spasticity; Gait Disorders, Neurologic | interventions — Botulinum Toxins, Type A

STUDY DESIGN:
Intervention Model Description: The design is a randomized controlled trial. One arm will be treated with a botulinum neurotoxin (BoTN) injection guided by the best available option, including ultrasonography + localized innervation zone (IZ) using anatomical references. The second arm will be treated with BoTN but guided with ultrasonography + in vivo location of the IZ using high-density electromyography.
Who Masked: Outcomes Assessor
Masking Description: The nature of the interventions makes blinding almost impossible. However, it will be possible to blind the support staff when they conduct the gait and functional evaluations. In the same way, the allocation of groups will be blinded at the time of performing the statistical analysis, which shall be performed by a third party.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Botulinum neurotoxin guided by ultrasonography and anatomical references (Active Comparator): Patients will be treated with a botulinum neurotoxin (BoNT) injection into the medial and lateral gastrocnemius muscles of the paretic hemi-body. This injection will be guided by ultrasonography and anatomical references described in the EUROMUSCULUS/USPRM guideline.
  Interventions: Combination Product: Botulinum toxin guided by ultrasonography and anatomical references
- Botulinum neurotoxin guided by ultrasonography and in vivo location of innervation zone (Experimental): Patients will be treated with a botulinum neurotoxin (BoNT) injection into the medial and lateral gastrocnemius muscles of the paretic hemi-body. However, in this case the injection will be guided by ultrasonography and the in vivo location of the innervation zones using noninvasive multielectrode electromyography.
  Interventions: Combination Product: Botulinum neurotoxin guided by ultrasonography and in vivo location of innervation zones guided by high-density electromyography

INTERVENTIONS:
Combination Product: Botulinum toxin guided by ultrasonography and anatomical references — The botulinum neurotoxin (BoNT) will be calculated according to the weight of each patient. It will be injected in four places: two of them into the medial gastrocnemius and the other two into the lateral gastrocnemius. For medial gastrocnemius muscle, ¼ of the dose will be injected into the muscle belly at the 25% of the distance between the popliteal fossa and the intermalleolar line. Another ¼ will be injected into the muscle belly at the 35% of the previously mentioned distance. For lateral gastrocnemius, ¼ of the dose will be injected into the muscle belly at the 20% of the distance between the popliteal fossa and the intermalleolar line. The remaining ¼ of the dose will be injected into the muscle belly at the 30% of the previously described distance. All patients will conduct the same physical therapy program and under the direction of the same team of physical therapists. This program will begin two weeks after receiving the BoNT injection.
  Other Names: Botox injection
  Arms: Botulinum neurotoxin guided by ultrasonography and anatomical references
Combination Product: Botulinum neurotoxin guided by ultrasonography and in vivo location of innervation zones guided by high-density electromyography — The botulinum neurotoxin (BoNT) will be calculated according to the weight of each patient. It will be injected in eight places: four will be located in vivo for gastrocnemius medialis and four for gastrocnemius lateralis. These places will correspond to innervation zones located by high-density electromyography in different zones of each muscle. Thus, each of the eight located innervation zones will receive 1/8 of the calculated dose for the gastrocnemius muscle. All patients will conduct the same physical therapy program and under the direction of the same team of physical therapists. This program will begin two weeks after receiving the BoNT injection.
  Other Names: Botox injection; Linear electrode array electromyography
  Arms: Botulinum neurotoxin guided by ultrasonography and in vivo location of innervation zone

SUMMARY:
According to our hypothesis, the use of HD-EMG shall allow an accurate localization of the innervations zones of the muscles, offering a better complement to the methodology applied so far to define the botulinum neurotoxin (BoNT) injection site. To achieve that goal, a randomized clinical trial comparing the effectiveness of two guiding methods to define the BoNT injection site in the gastrocnemius muscles will be conducted. One arm will be guided with ultrasonography + localized IZ using anatomical references; while the second arm with ultrasonography + in vivo location of the IZ through HD-EMG. The effectiveness will be evaluated by changes in functional tests and in biomechanical parameters of the gait assessed with a three-dimensional motion analysis system. These outcomes will be measured at baseline (T0), at three (T3w) and six weeks (T6w), post BoNT injection. The differences between sessions will be evaluated as measurements of effectiveness. We expect that greater effectiveness will be found in the group that receives the injection of BoNT, guided by the in vivo location of the IZ.

DETAILED DESCRIPTION:
This research proposal seeks to improve the current procedures to determinate the botulinum neurotoxin (BoNT) injection site. More precisely, we propose to complement the ultrasonography with an in vivo location of the IZ, using a non-invasive technique based on surface multielectrode electromyography grid, which is called high density-surface EMG (HD-EMG). According to our hypothesis, the use of HD-EMG shall allow an accurate localization of the IZs of the muscles, offering a better complement to the methodology applied so far to define the BoNT injection site. To achieve that goal, a randomized clinical trial comparing the effectiveness of two guiding methods to define the BoNT injection site in the gastrocnemius muscles (main ankle extensors or plantar flexors) will be conducted. One arm will be treated with the best available option, which includes ultrasonography + localized IZ using anatomical references. The second arm will be managed using ultrasonography + in vivo location of the IZ through. The last will be measured using HD-EMG by recording the motor unit action potentials along the muscle fibers. This technique can identify the location of the IZ by the change of phase of those potentials. The effectiveness will be evaluated by changes in biomechanical parameters of the gait, assessed using a three-dimensional motion analysis system. The outcomes will be biomechanical gait variables associated with the ankle joint (ankle joint moment, dorsiflexion range, among others) and functional tests (spasticity using Ashworth scale, 6-minute walk test and the Timed Up and Go Test). These outcomes will be evaluated at baseline (T0), at three (T3w) and six weeks (T6w), post BoNT injection. The differences between sessions will be evaluated as measurements of effectiveness (Delta1 = T3w-T0; Delta2 = T6w - T0). To compare the effectiveness between groups, these delta values will be compared using a student's t-test or a Mann-Whitney U test, as appropriate. Also, a Cohen's d will be calculated to determine the magnitude of these differences. In addition, the post-hoc power (1-β) will be measured. All statistical analyses will be performed in the STATA software (version 14.0 Stata-Corp LP, USA), considering a one tailed analysis, and a confidence level of 95%. Statistically significant differences will be considered those associated with a p-value lower than 0.05. We expect to find greater effectiveness in the group that receives the injection of BoNT, guided by the in vivo location of the IZ using HD-EMG.

ELIGIBILITY:
Inclusion Criteria:

* Hemiplegia secondary to an ischemic of hemorrhagic stroke.
* Focal spasticity of gastrocnemius muscles status 1-3 according to the modified Ashworth scale.
* Independent gait ability with or without the use of technical assistance.

Exclusion Criteria:

* Spasticity status 4 according to the modified Ashworth scale.
* Focal spasticity of the tibialis posterior and/or soleus.
* Fracture and/or contracture in the lower extremities.
* Other medical treatment for spasticity.
* Allergy to the botulinum neurotoxin.
* Suffering from some infectious disease
* Pregnancy or breastfeeding

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 18 (Actual)
Dates: Start 2022-07-01 (Actual); Primary Completion 2022-11-29 (Actual); Study Completion 2022-12-04 (Actual)

PRIMARY OUTCOMES:
Maximum ankle dorsiflexion during the stance phase in the paretic limb. | Before intervention (T0), three weeks (T3w) and six weeks (T6w) post botulinum neurotoxin injection
  Peak dorsiflexion angle during the stance phase in the paretic limb. This value will be calculated from Vicon Nexus 2.12 software, using the conventional gait model + functional calibration, and will be considered as the average value within 8 to 10 gait cycles.
Maximum ankle plantarflexion moment during the stance phase in the paretic limb | Before intervention (T0), three weeks (T3w) and six weeks (T6w) post botulinum neurotoxin injection.
  Peak internal ankle dorsiflexion moment during the stance phase in the paretic limb. This value will be calculated from Vicon Nexus 2.12 software, using the conventional gait model + functional calibration, and will be considered as the average value within 8 to 10 gait cycles.
Foot clearance in the paretic limb. | Before intervention (T0), three weeks (T3w) and six weeks (T6w) post botulinum neurotoxin injection.
  Minimum distance between the lowest point on the shoe and the ground during the swing phase in the paretic limb. This value will be calculated from a custom-made biomechanical model, and will be considered as the average value within 8 to 10 gait cycles.

SECONDARY OUTCOMES:
Spasticity of plantar flexor muscles using the Ashworth modified scale. | Before intervention (T0), three weeks (T3w) and six weeks (T6w) post botulinum neurotoxin injection.
  Qualitative evaluation of the increase in ankle plantar flexors tone during a muscle stretch movement (dorsiflexion). This will be scaled from 0 (no increase in muscle tone) to 4 (ankle rigid during dorsiflexion movement).
6-minute walk distance. | Before intervention (T0), three weeks (T3w) and six weeks (T6w) post botulinum neurotoxin injection.
  Measurement of distance walked over a span of 6 minutes.
Timed up and go time. | Before intervention (T0), three weeks (T3w) and six weeks (T6w) post botulinum neurotoxin injection.
  Time to complete a standing from a chair with no arms, walking 5 meters and returning to sit down.

CONTACTS AND LOCATIONS:
Overall Officials: Rodrigo A Guzmán-Venegas, PhD, Study Director — Universidad de los Andes, Chile
Locations (2):
- Chile (2):
  - Universidad de los Andes, Santiago, Las Condes
  - Instituto Nacional de Rehabilitación Pedro Aguirre Cerda, Santiago, Peñalolen

IPD SHARING:
Plan to Share IPD: Yes
Study protocol and statistical analysis plan will be published. Statistical analysis plan includes all databases used in the study. These databases will not include personal information of patients.
Supporting Information: Study Protocol, SAP
Time Frame: Previously mentioned data will be available 6 months after publication.
Access Criteria: For access to research data, researchers must send a "data access statement" to the principal investigator (Rodrigo Guzmán-Venegas, rguzman@uandes.cl). This request must include as much information as possible about the use of the data. Also, it must include contact information (telephone number and e-mail to contact) on the petitioner.

REFERENCES:
- [Background] Grysiewicz RA, Thomas K, Pandey DK. Epidemiology of ischemic and hemorrhagic stroke: incidence, prevalence, mortality, and risk factors. Neurol Clin. 2008 Nov;26(4):871-95, vii. doi: 10.1016/j.ncl.2008.07.003. PMID 19026895
- [Background] Lavados PM, Sacks C, Prina L, Escobar A, Tossi C, Araya F, Feuerhake W, Galvez M, Salinas R, Alvarez G. Incidence, 30-day case-fatality rate, and prognosis of stroke in Iquique, Chile: a 2-year community-based prospective study (PISCIS project). Lancet. 2005 Jun 25-Jul 1;365(9478):2206-15. doi: 10.1016/S0140-6736(05)66779-7. PMID 15978929
- [Background] Watkins CL, Leathley MJ, Gregson JM, Moore AP, Smith TL, Sharma AK. Prevalence of spasticity post stroke. Clin Rehabil. 2002 Aug;16(5):515-22. doi: 10.1191/0269215502cr512oa. PMID 12194622
- [Background] von Schroeder HP, Coutts RD, Lyden PD, Billings E Jr, Nickel VL. Gait parameters following stroke: a practical assessment. J Rehabil Res Dev. 1995 Feb;32(1):25-31. PMID 7760264
- [Background] Dashtipour K, Chen JJ, Walker HW, Lee MY. Systematic Literature Review of AbobotulinumtoxinA in Clinical Trials for Lower Limb Spasticity. Medicine (Baltimore). 2016 Jan;95(2):e2468. doi: 10.1097/MD.0000000000002468. PMID 26765447
- [Background] Wei TS, Liu PT, Chang LW, Liu SY. Gait asymmetry, ankle spasticity, and depression as independent predictors of falls in ambulatory stroke patients. PLoS One. 2017 May 23;12(5):e0177136. doi: 10.1371/journal.pone.0177136. eCollection 2017. PMID 28542281
- [Background] Lance JW. The control of muscle tone, reflexes, and movement: Robert Wartenberg Lecture. Neurology. 1980 Dec;30(12):1303-13. doi: 10.1212/wnl.30.12.1303. No abstract available. PMID 7192811
- [Background] Schroder AS, Fietzek UM, Pavicic T, Stehr M, Baumann AC, Ruzicka T, Heinen F. [Botulinum toxin--the all-rounder in medicine]. MMW Fortschr Med. 2011 Jan 27;153(4):33-9; quiz 40. doi: 10.1007/BF03367697. No abstract available. German. PMID 22165615
- [Background] Woolley SM. Characteristics of gait in hemiplegia. Top Stroke Rehabil. 2001 Winter;7(4):1-18. doi: 10.1310/JB16-V04F-JAL5-H1UV. PMID 14523755
- [Background] Cofre Lizama LE, Khan F, Galea MP. Beyond speed: Gait changes after botulinum toxin injections in chronic stroke survivors (a systematic review). Gait Posture. 2019 May;70:389-396. doi: 10.1016/j.gaitpost.2019.03.035. Epub 2019 Apr 4. PMID 30974394
- [Background] Karadag-Saygi E, Cubukcu-Aydoseli K, Kablan N, Ofluoglu D. The role of kinesiotaping combined with botulinum toxin to reduce plantar flexors spasticity after stroke. Top Stroke Rehabil. 2010 Jul-Aug;17(4):318-22. doi: 10.1310/tsr1704-318. PMID 20826420
- [Background] Hesse S, Krajnik J, Luecke D, Jahnke MT, Gregoric M, Mauritz KH. Ankle muscle activity before and after botulinum toxin therapy for lower limb extensor spasticity in chronic hemiparetic patients. Stroke. 1996 Mar;27(3):455-60. doi: 10.1161/01.str.27.3.455. PMID 8610313
- [Background] Pradon D, Hutin E, Khadir S, Taiar R, Genet F, Roche N. A pilot study to investigate the combined use of Botulinum toxin type-a and ankle foot orthosis for the treatment of spastic foot in chronic hemiplegic patients. Clin Biomech (Bristol). 2011 Oct;26(8):867-72. doi: 10.1016/j.clinbiomech.2011.04.003. Epub 2011 May 17. PMID 21592635
- [Background] Castelao M, Marques RE, Duarte GS, Rodrigues FB, Ferreira J, Sampaio C, Moore AP, Costa J. Botulinum toxin type A therapy for cervical dystonia. Cochrane Database Syst Rev. 2017 Dec 12;12(12):CD003633. doi: 10.1002/14651858.CD003633.pub3. PMID 29230798
- [Background] Borodic G. Therapeutic botulinum toxin. Lancet. 1994 Nov 12;344(8933):1370. doi: 10.1016/s0140-6736(94)90732-3. No abstract available. PMID 7968058
- [Background] Kaymak B, Kara M, Yagiz On A, Soylu AR, Ozcakar L. Innervation zone targeted botulinum toxin injections. Eur J Phys Rehabil Med. 2018 Feb;54(1):100-109. doi: 10.23736/S1973-9087.17.04663-9. Epub 2017 Mar 6. PMID 28264545
- [Background] Lapatki BG, van Dijk JP, van de Warrenburg BP, Zwarts MJ. Botulinum toxin has an increased effect when targeted toward the muscle's endplate zone: a high-density surface EMG guided study. Clin Neurophysiol. 2011 Aug;122(8):1611-6. doi: 10.1016/j.clinph.2010.11.018. Epub 2010 Dec 30. PMID 21195024
- [Background] Delnooz CC, Veugen LC, Pasman JW, Lapatki BG, van Dijk JP, van de Warrenburg BP. The clinical utility of botulinum toxin injections targeted at the motor endplate zone in cervical dystonia. Eur J Neurol. 2014 Dec;21(12):1486-e98. doi: 10.1111/ene.12517. Epub 2014 Jul 24. PMID 25060697
- [Background] Mirelman A, Shema S, Maidan I, Hausdorff JM. Gait. Handb Clin Neurol. 2018;159:119-134. doi: 10.1016/B978-0-444-63916-5.00007-0. PMID 30482309
- [Background] Fugl-Meyer AR, Jaasko L, Norlin V. The post-stroke hemiplegic patient. II. Incidence, mortality, and vocational return in Goteborg, Sweden with a review of the literature. Scand J Rehabil Med. 1975;7(2):73-83. PMID 1162302
- [Background] Beyaert C, Vasa R, Frykberg GE. Gait post-stroke: Pathophysiology and rehabilitation strategies. Neurophysiol Clin. 2015 Nov;45(4-5):335-55. doi: 10.1016/j.neucli.2015.09.005. Epub 2015 Nov 4. PMID 26547547
- [Background] Mahendran N, Kuys SS, Brauer SG. Recovery of ambulation activity across the first six months post-stroke. Gait Posture. 2016 Sep;49:271-276. doi: 10.1016/j.gaitpost.2016.06.038. Epub 2016 Jun 29. PMID 27474947
- [Background] Winter DA. Overall principle of lower limb support during stance phase of gait. J Biomech. 1980;13(11):923-7. doi: 10.1016/0021-9290(80)90162-1. No abstract available. PMID 7275999
- [Background] Kaymak B, Kara M, Tok F, Ulasli AM, Ozturk GT, Chang KV, Hsiao MY, Hung CY, Yagiz On A, Ozcakar L. Sonographic guide for botulinum toxin injections of the lower limb: EUROMUSCULUS/USPRM spasticity approach. Eur J Phys Rehabil Med. 2018 Jun;54(3):486-498. doi: 10.23736/S1973-9087.17.04667-6. Epub 2017 Apr 4. PMID 28382814
- [Background] Akturk S, Buyukavci R, Ersoy Y. Functional outcomes following ultrasound-guided botulinum toxin type A injections to reduce spastic equinovarus in adult post-stroke patients. Toxicon. 2018 May;146:95-98. doi: 10.1016/j.toxicon.2018.03.003. Epub 2018 Mar 9. PMID 29530514
- [Background] Kwon JY, Hwang JH, Kim JS. Botulinum toxin a injection into calf muscles for treatment of spastic equinus in cerebral palsy: a controlled trial comparing sonography and electric stimulation-guided injection techniques: a preliminary report. Am J Phys Med Rehabil. 2010 Apr;89(4):279-86. doi: 10.1097/PHM.0b013e3181ca24ac. PMID 20068435
- [Background] Park GY, Kwon DR. Sonoelastographic evaluation of medial gastrocnemius muscles intrinsic stiffness after rehabilitation therapy with botulinum toxin a injection in spastic cerebral palsy. Arch Phys Med Rehabil. 2012 Nov;93(11):2085-9. doi: 10.1016/j.apmr.2012.06.024. Epub 2012 Jul 7. PMID 22776155
- [Background] Picelli A, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Tamburin S, Girardi P, Gimigliano R, Smania N. Accuracy of botulinum toxin type A injection into the gastrocnemius muscle of adults with spastic equinus: manual needle placement and electrical stimulation guidance compared using ultrasonography. J Rehabil Med. 2012 May;44(5):450-2. doi: 10.2340/16501977-0970. PMID 22549655
- [Background] Picelli A, Tamburin S, Bonetti P, Fontana C, Barausse M, Dambruoso F, Gajofatto F, Santilli V, Smania N. Botulinum toxin type A injection into the gastrocnemius muscle for spastic equinus in adults with stroke: a randomized controlled trial comparing manual needle placement, electrical stimulation and ultrasonography-guided injection techniques. Am J Phys Med Rehabil. 2012 Nov;91(11):957-64. doi: 10.1097/PHM.0b013e318269d7f3. PMID 23085706
- [Background] Amatya B, Cofre Lizama LE, Elmalik A, Bastani A, Galea MP, Khan F. Multidimensional evaluation of changes in limb function following botulinum toxin injection in persons with stroke. NeuroRehabilitation. 2019;45(1):67-78. doi: 10.3233/NRE-192722. PMID 31403954
- [Background] Masuda T, Miyano H, Sadoyama T. The propagation of motor unit action potential and the location of neuromuscular junction investigated by surface electrode arrays. Electroencephalogr Clin Neurophysiol. 1983 May;55(5):594-600. doi: 10.1016/0013-4694(83)90171-2. PMID 6187554
- [Background] Tokunaga T, Baba S, Tanaka M, Kashiwagi K, Kimura K, Kawazoe T. Two-dimensional configuration of the myoneural junctions of human masticatory muscle detected with matrix electrode. J Oral Rehabil. 1998 May;25(5):329-34. doi: 10.1046/j.1365-2842.1998.00199.x. PMID 9639155
- [Background] Masuda T, Sadoyama T. Topographical map of innervation zones within single motor units measured with a grid surface electrode. IEEE Trans Biomed Eng. 1988 Aug;35(8):623-8. doi: 10.1109/10.4595. No abstract available. PMID 3169813
- [Background] Masuda T, Sadoyama T. Distribution of innervation zones in the human biceps brachii. J Electromyogr Kinesiol. 1991 Jun;1(2):107-15. doi: 10.1016/1050-6411(91)90004-O. PMID 20870500
- [Background] Saitou K, Masuda T, Michikami D, Kojima R, Okada M. Innervation zones of the upper and lower limb muscles estimated by using multichannel surface EMG. J Hum Ergol (Tokyo). 2000 Dec;29(1-2):35-52. PMID 12696320
- [Background] Van Campenhout A, Hubens G, Fagard K, Molenaers G. Localization of motor nerve branches of the human psoas muscle. Muscle Nerve. 2010 Aug;42(2):202-7. doi: 10.1002/mus.21660. PMID 20544927
- [Background] Yu DZ, Liu AT, Dang RS, Zhang CS, Zhang JL, Chen G, Yi J, Han T, Jiang H. Intramuscular innervations of muscle flaps that are commonly used in clinical settings. Surg Radiol Anat. 2010 Aug;32(7):637-46. doi: 10.1007/s00276-010-0644-2. Epub 2010 Mar 13. PMID 20229172
- [Background] Kwon JY, Kim JS, Lee WI. Anatomic localization of motor points of hip adductors. Am J Phys Med Rehabil. 2009 Apr;88(4):336-41. doi: 10.1097/PHM.0b013e3181619435. PMID 18174845
- [Background] Crystal R, Malone AA, Eastwood DM. Motor points for neuromuscular blockade of the adductor muscle group. Clin Orthop Relat Res. 2005 Aug;(437):196-200. doi: 10.1097/01.blo.0000165856.38166.9a. PMID 16056049
- [Background] Won SY, Rha DW, Kim HS, Jung SH, Park ES, Hu KS, Kim HJ. Intramuscular nerve distribution pattern of the adductor longus and gracilis muscles demonstrated with Sihler staining: guidance for botulinum toxin injection. Muscle Nerve. 2012 Jul;46(1):80-5. doi: 10.1002/mus.23273. Epub 2012 May 29. PMID 22644785
- [Background] Kumar VP, Liu J, Lau HK, Pereira BP, Shen Y, Pho RW. Neurovascular supply of the gracilis muscle: a study in the monkey and human. Plast Reconstr Surg. 1998 Jun;101(7):1854-60. doi: 10.1097/00006534-199806000-00012. PMID 9623827
- [Background] Paul AC. Muscle length affects the architecture and pattern of innervation differently in leg muscles of mouse, guinea pig, and rabbit compared to those of human and monkey muscles. Anat Rec. 2001 Mar 1;262(3):301-9. doi: 10.1002/1097-0185(20010301)262:33.0.CO;2-H. PMID 11241198
- [Background] BUCHTHAL F, GULD C, ROSENFALCK P. Action potential parameters in normal human muscle and their dependence on physical variables. Acta Physiol Scand. 1954 Nov;32(2-3):200-18. doi: 10.1111/j.1748-1716.1954.tb01167.x. No abstract available. PMID 13228109
- [Background] BUCHTHAL F, GULD C, ROSENFALCK P. Innervation zone and propagation velocity in human muscle. Acta Physiol Scand. 1955 Dec 31;35(2):174-90. doi: 10.1111/j.1748-1716.1955.tb01276.x. No abstract available. PMID 13301862
- [Background] Buchthal F. Spontaneous electrical activity: an overview. Muscle Nerve. 1982;5(9S):S52-9. PMID 6763149
- [Background] Childers MK. The importance of electromyographic guidance and electrical stimulation for injection of botulinum toxin. Phys Med Rehabil Clin N Am. 2003 Nov;14(4):781-92. doi: 10.1016/s1047-9651(03)00047-0. PMID 14580037
- [Background] Childers MK. Targeting the neuromuscular junction in skeletal muscles. Am J Phys Med Rehabil. 2004 Oct;83(10 Suppl):S38-44. doi: 10.1097/01.phm.0000141129.23219.42. PMID 15448576
- [Background] Castroflorio T, Farina D, Bottin A, Debernardi C, Bracco P, Merletti R, Anastasi G, Bramanti P. Non-invasive assessment of motor unit anatomy in jaw-elevator muscles. J Oral Rehabil. 2005 Oct;32(10):708-13. doi: 10.1111/j.1365-2842.2005.01490.x. PMID 16159347
- [Background] Merletti R, Farina D, Gazzoni M. The linear electrode array: a useful tool with many applications. J Electromyogr Kinesiol. 2003 Feb;13(1):37-47. doi: 10.1016/s1050-6411(02)00082-2. PMID 12488085
- [Background] Ullah K, Cescon C, Afsharipour B, Merletti R. Automatic detection of motor unit innervation zones of the external anal sphincter by multichannel surface EMG. J Electromyogr Kinesiol. 2014 Dec;24(6):860-7. doi: 10.1016/j.jelekin.2014.05.003. Epub 2014 May 24. PMID 24948528
- [Background] Guzman-Venegas RA, Bralic MP, Cordero JJ, Cavada G, Araneda OF. Concordance of the location of the innervation zone of the tibialis anterior muscle using voluntary and imposed contractions by electrostimulation. J Electromyogr Kinesiol. 2016 Apr;27:18-23. doi: 10.1016/j.jelekin.2016.01.002. Epub 2016 Jan 29. PMID 26874077
- [Background] Kara M, Kaymak B, Ulasli AM, Tok F, Ozturk GT, Chang KV, Hsiao MY, Hung CY, Yagiz On A, Ozcakar L. Sonographic guide for botulinum toxin injections of the upper limb: EUROMUSCULUS/USPRM spasticity approach. Eur J Phys Rehabil Med. 2018 Jun;54(3):469-485. doi: 10.23736/S1973-9087.17.04664-0. Epub 2017 Mar 6. PMID 28264546
- [Background] Lim EC, Seet RC. Botulinum toxin: description of injection techniques and examination of controversies surrounding toxin diffusion. Acta Neurol Scand. 2008 Feb;117(2):73-84. doi: 10.1111/j.1600-0404.2007.00931.x. Epub 2007 Sep 11. PMID 17850405
- [Background] Lee JH, Han SH, Ye JF, Lee BN, An X, Kwon SO. Effective zone of botulinum toxin a injections in hallux claw toe syndrome: an anatomical study. Muscle Nerve. 2012 Feb;45(2):217-21. doi: 10.1002/mus.22263. PMID 22246877
- [Background] Lee DR, You JH, Yi CH, Jeon HS. Motor point location index using regression equations for the tibialis anterior muscle. NeuroRehabilitation. 2012;30(4):307-13. doi: 10.3233/NRE-2012-0760. PMID 22672945
- [Background] Guzman-Venegas RA, Araneda OF, Silvestre RA. Differences between motor point and innervation zone locations in the biceps brachii. An exploratory consideration for the treatment of spasticity with botulinum toxin. J Electromyogr Kinesiol. 2014 Dec;24(6):923-7. doi: 10.1016/j.jelekin.2014.07.012. Epub 2014 Aug 2. PMID 25138645
- [Background] Nishizono H, Saito Y, Miyashita M. The estimation of conduction velocity in human skeletal muscle in situ with surface electrodes. Electroencephalogr Clin Neurophysiol. 1979 Jun;46(6):659-64. doi: 10.1016/0013-4694(79)90103-2. PMID 87310
- [Background] Grigoriu AI, Dinomais M, Remy-Neris O, Brochard S. Impact of Injection-Guiding Techniques on the Effectiveness of Botulinum Toxin for the Treatment of Focal Spasticity and Dystonia: A Systematic Review. Arch Phys Med Rehabil. 2015 Nov;96(11):2067-78.e1. doi: 10.1016/j.apmr.2015.05.002. Epub 2015 May 14. PMID 25982240
- [Background] Meseguer-Henarejos AB, Sanchez-Meca J, Lopez-Pina JA, Carles-Hernandez R. Inter- and intra-rater reliability of the Modified Ashworth Scale: a systematic review and meta-analysis. Eur J Phys Rehabil Med. 2018 Aug;54(4):576-590. doi: 10.23736/S1973-9087.17.04796-7. Epub 2017 Sep 13. PMID 28901119
- [Background] Clague-Baker N, Robinson T, Hagenberg A, Drewry S, Gillies C, Singh S. The validity and reliability of the Incremental Shuttle Walk Test and Six-minute Walk Test compared to an Incremental Cycle Test for people who have had a mild-to-moderate stroke. Physiotherapy. 2019 Jun;105(2):275-282. doi: 10.1016/j.physio.2018.12.005. Epub 2018 Dec 21. PMID 30954276
- [Background] Geiger M, Bonnyaud C, Bussel B, Roche N. Assessing of imagined and real expanded Timed Up and Go tests in patients with chronic stroke: A case-control study. J Rehabil Med. 2018 May 8;50(5):413-419. doi: 10.2340/16501977-2315. PMID 29487942
- [Background] Comella CL, Buchman AS, Tanner CM, Brown-Toms NC, Goetz CG. Botulinum toxin injection for spasmodic torticollis: increased magnitude of benefit with electromyographic assistance. Neurology. 1992 Apr;42(4):878-82. doi: 10.1212/wnl.42.4.878. PMID 1565246
- [Background] Kaishou Xu, Tiebin Yan, Jianning Mai. A randomized controlled trial to compare two botulinum toxin injection techniques on the functional improvement of the leg of children with cerebral palsy. Clin Rehabil. 2009 Sep;23(9):800-11. doi: 10.1177/0269215509335295. Epub 2009 May 29. PMID 19482892
- [Background] Jordan SE, Ahn SS, Gelabert HA. Combining ultrasonography and electromyography for botulinum chemodenervation treatment of thoracic outlet syndrome: comparison with fluoroscopy and electromyography guidance. Pain Physician. 2007 Jul;10(4):541-6. PMID 17660852
- [Background] Gracies JM, Lugassy M, Weisz DJ, Vecchio M, Flanagan S, Simpson DM. Botulinum toxin dilution and endplate targeting in spasticity: a double-blind controlled study. Arch Phys Med Rehabil. 2009 Jan;90(1):9-16.e2. doi: 10.1016/j.apmr.2008.04.030. PMID 19154823
- [Background] Kaymak B, Kara M, Gurcay E, Ozcakar L. Sonographic Guide for Botulinum Toxin Injections of the Neck Muscles in Cervical Dystonia. Phys Med Rehabil Clin N Am. 2018 Feb;29(1):105-123. doi: 10.1016/j.pmr.2017.08.009. PMID 29173657
- [Background] Rohrig B, du Prel JB, Wachtlin D, Blettner M. Types of study in medical research: part 3 of a series on evaluation of scientific publications. Dtsch Arztebl Int. 2009 Apr;106(15):262-8. doi: 10.3238/arztebl.2009.0262. Epub 2009 Apr 10. PMID 19547627
- [Background] Paterson KL, Hinman RS, Metcalf BR, Bennell KL, Wrigley TV. Plug-in-Gait calculation of the knee adduction moment in people with knee osteoarthritis during shod walking: comparison of two different foot marker models. J Foot Ankle Res. 2017 Feb 4;10:8. doi: 10.1186/s13047-017-0187-4. eCollection 2017. PMID 28174605
- [Background] Lin LI. A concordance correlation coefficient to evaluate reproducibility. Biometrics. 1989 Mar;45(1):255-68. PMID 2720055
- [Background] Bland JM, Altman DG. Statistical methods for assessing agreement between two methods of clinical measurement. Lancet. 1986 Feb 8;1(8476):307-10. PMID 2868172
- [Background] Sullivan GM, Feinn R. Using Effect Size-or Why the P Value Is Not Enough. J Grad Med Educ. 2012 Sep;4(3):279-82. doi: 10.4300/JGME-D-12-00156.1. No abstract available. PMID 23997866